CLINICAL TRIAL: NCT00871351
Title: Ezetimibe Phase IV Clinical Study in Patients With Hypercholesterolemia
Brief Title: Evaluation of Ezetimibe and Atorvastatin Coadministration Versus Atorvastatin or Rosuvastatin Monotherapy in Japanese Patients With Hypercholesterolemia (Study P06027)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P06027
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Results first posted 2011-08-23 (Estimated); Last update posted 2024-05-23 (Actual); Status verified 2022-02

CONDITIONS: Primary Hypercholesterolemia
MeSH Terms: interventions — Ezetimibe; Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ezetimibe + Atorvastatin (Experimental): Participants with hypercholesterolemia receiving atorvastatin 10 mg and ezetimibe 10 mg for 12 weeks after a 4-week washout and 4 weeks of daily atorvastatin 10 mg
  Interventions: Drug: Ezetimibe; Drug: Atorvastatin
- Atorvastatin (Active Comparator): Participants with hypercholesterolemia receiving atorvastatin 20 mg for 12 weeks after a 4-week washout and 4 weeks of daily atorvastatin 10 mg
  Interventions: Drug: Atorvastatin
- Rosuvastatin (Active Comparator): Participants with hypercholesterolemia receiving rosuvastatin 2.5 mg for 12 weeks after a 4-week washout and 4 weeks of daily atorvastatin 10 mg
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Ezetimibe — 1 tablet of 10 mg daily for 12 weeks (Weeks 5-16)
  Other Names: SCH 058235
  Arms: Ezetimibe + Atorvastatin
Drug: Atorvastatin — 1 tablet of 10 mg daily for 12 weeks (Weeks 5-16)
  Arms: Ezetimibe + Atorvastatin
Drug: Atorvastatin — 2 tablets of 10 mg daily for 12 weeks (Weeks 5-16)
  Arms: Atorvastatin
Drug: Rosuvastatin — 1 tablet of 2.5 mg daily for 12 weeks (Weeks 5-16)
  Arms: Rosuvastatin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of atorvastatin 10 mg and ezetimibe 10 mg coadministration in Japanese participants with hypercholesterolemia whose low-density lipoprotein (LDL)-cholesterol levels have not reached the lipid management target value with atorvastatin 10 mg alone, versus increasing the dose of atorvastatin to 20 mg or changing to rosuvastatin 2.5 mg.

ELIGIBILITY:
Inclusion Criteria:

* atorvastatin 10 mg monotherapy for 4 weeks or longer before the start of the 4-week washout and low density lipoprotein-cholesterol (LDL-C) levels that had not reached the following lipid management target values during treatment: Category I (low-risk group) with no other risk factors - LDL-C <160 mg/dL; Category II (mid-risk group) with 1-2 risk factors other than LDL-C levels - LDL-C <140 mg/dL; Category III (high-risk group) with 3 or more other risk factors - LDL-C <120 mg/dL; and for participants with history of coronary artery disease - LDL-C <100 mg/dL.
* outpatient men or women, age 20 years and older

Exclusion Criteria:

* fasted triglyceride level at the start of washout or treatment period exceeding 400 mg/dL.
* homozygous familial hypercholesterolemia.
* creatine phosphokinase (CPK) >2 times the upper limit of normal (X ULN) at start of washout or treatment period.
* glycosylated hemoglobin (HbA1c) >=8％ at start of washout or treatment period.
* severe hepatic function disorder, or aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2X ULN at start of washout or treatment period.
* hypersensitivity to ezetimibe, atorvastatin, or rosuvastatin tablets.
* pregnant or lactating
* discontinued use of atorvastatin 10 mg for less than 4 weeks at start of treatment period (however, if participant had taken atorvastatin 10 mg before the test conducted at the start of the observation period, a period of discontinuation of 27 days is allowed.)
* cyclosporine treatment
* hyperlipidemia associated with hypothyroidism, obstructive gall bladder or biliary disease, chronic renal failure, and/or pancreatitis.
* hyperlipidemia associated with drug administration that causes adverse serum lipid effects.
* participation in a clinical study within 4 weeks of washout
* cancer or cancer history within previous 5 years, except for successfully treated basal cell carcinoma of the skin.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2009-02-01 (Actual); Primary Completion 2010-05-01 (Actual); Study Completion 2010-05-01 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Teramoto T, Sawada T, Iwamoto K, Daida H. Clinical Efficacy and Tolerability of Ezetimibe in Combination With Atorvastatin in Japanese Patients With Hypercholesterolemia-Ezetimibe Phase IV Randomized Controlled Trial in Patients With Hypercholesterolemia. Curr Ther Res Clin Exp. 2012 Feb;73(1-2):16-40. doi: 10.1016/j.curtheres.2012.02.002. PMID 24653510

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ezetimibe + Atorvastatin | Atorvastatin | Rosuvastatin
Started | 47 | 46 | 32
Completed | 43 | 45 | 32
Not Completed | 4 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Adverse Event | 3 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ezetimibe + Atorvastatin | Atorvastatin | Rosuvastatin | Total
Number analyzed (Participants) | 47 | 46 | 32 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (11.4) | 59.3 (11.8) | 61.1 (12.0) | 61.0 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 22 | 17 | 64
  Male | 22 | 24 | 15 | 61
Region of Enrollment [Number; unit: participants]
  Japan | 47 | 46 | 32 | 125

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Low-Density Lipoprotein - Cholesterol (LDL-C) Values
Description: LDL-C was measured before group study drug administration (Week 4, end of atorvastatin single therapy) and at the end of study drug administration (after 12 weeks of study drug treatment, or at discontinuation).
Time Frame: End of Week 4 to Week 16 or discontinuation
Population: Randomized participants
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Ezetimibe + Atorvastatin | Atorvastatin | Rosuvastatin
Number analyzed (Participants) | 47 | 46 | 32
Percent change | -25.8 [-29.2 to -22.4] | -15.1 [-18.6 to -11.7] | 0.8 [-3.3 to 4.9]
Statistical Analysis 1: Comparison: Ezetimibe + Atorvastatin vs Atorvastatin; Test type: Superiority or Other; p < 0.0001, Hochberg's method; Mean Difference (Net) = -10.6, 95% CI 2-sided [-15.4 to -5.8]
Statistical Analysis 2: Comparison: Ezetimibe + Atorvastatin vs Rosuvastatin; Test type: Superiority or Other; p < 0.0001, Hochberg's method; Mean Difference (Net) = -26.5, 95% CI 2-sided [-31.8 to -21.2]

2. Secondary Outcome: Percent Change in LDL-C
Description: LDL-C was measured at the start of the atorvastatin 10 mg treatment period (end of the washout period) and at the end of administration of the study drug (Week 16 or discontinuation).
Time Frame: End of washout period to Week 16 or discontinuation
Population: Randomized participants
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Ezetimibe + Atorvastatin | Atorvastatin | Rosuvastatin
Number analyzed (Participants) | 47 | 46 | 32
Percent change | -49.6 [-52.9 to -46.4] | -41.1 [-44.4 to -37.9] | -30.5 [-34.4 to -26.6]
Statistical Analysis 1: Comparison: Ezetimibe + Atorvastatin vs Atorvastatin; Test type: Superiority or Other; p = 0.0003, Hochberg's method
Statistical Analysis 2: Comparison: Ezetimibe + Atorvastatin vs Rosuvastatin; Test type: Superiority or Other; p < 0.0001, Hochberg's method

3. Secondary Outcome: Number of Participants Whose LDL-C Levels Reached the Lipid Management Target Values
Description: LDL-C was measured at the end of administration of the study drug (Week 16 or discontinuation).
  Target values:
  For participants with history of coronary artery disease: <100 mg/dL;
  for participants with at least 3 cardiovascular (CV) risk factors: <120 mg/dL;
  for participants with 1-2 CV risk factors: <140 mg/dL;
  for participants with no CV risk factors: <160 mg/dL.
Time Frame: Week 16 or discontinuation
Population: Randomized participants
Measure: Number; unit: Participants
Arm/Group | Ezetimibe + Atorvastatin | Atorvastatin | Rosuvastatin
Number analyzed (Participants) | 47 | 46 | 32
Participants | 37 | 19 | 1

4. Secondary Outcome: Percent Change in Total Lipids and High Sensitivity C-reactive Protein (Hs-CRP)
Description: Total cholesterol, triglycerides, high-density lipoprotein cholesterol (HDL-C), non-HDL-C, and hs-CRP were measured at 4 weeks after the start of the treatment period (after completion of administration of atorvastatin 10 mg alone) and at Week 16 or at discontinuation.
Time Frame: End of Week 4 to Week 16 or discontinuation
Population: Randomized participants
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Ezetimibe + Atorvastatin | Atorvastatin | Rosuvastatin
Number analyzed (Participants) | 47 | 46 | 32
Percent change
  Total Cholesterol | -18.0 [-20.7 to -15.2] | -10.3 [-13.1 to -7.4] | 1.9 [-1.7 to 5.5]
  Triglycerides | -0.8 [-14.4 to 12.8] | 0.2 [-10.9 to 11.4] | 14.7 [2.3 to 27.0]
  High-Density Lipoprotein Cholesterol (HDL-C) | 4.5 [0.9 to 8.2] | 0.5 [-2.6 to 3.5] | 2.5 [-1.4 to 6.4]
  Non-HDL-C | -25.0 [-28.5 to -21.5] | -13.7 [-17.0 to -10.3] | 2.0 [-2.6 to 6.5]
  High Sensitivity C-Reactive Protein (Hs-CRP) | 49.0 [-43.2 to 141.3] | 9.9 [-24.1 to 43.9] | 25.7 [-4.8 to 56.1]

5. Secondary Outcome: Percent Change in Total Lipids and Hs-CRP
Description: Total cholesterol, triglycerides, high-density lipoprotein cholesterol (HDL-C), non-HDL-C, and hs-CRP were measured at the start of the treatment period (at start of administration of atorvastatin 10 mg alone) and at the end of study drug (Week 16 or discontinuation).
Time Frame: End of washout to Week 16 or discontinuation
Population: Randomized participants
Measure: Mean (95% Confidence Interval); unit: Percent change
Arm/Group | Ezetimibe + Atorvastatin | Atorvastatin | Rosuvastatin
Number analyzed (Participants) | 47 | 46 | 32
Percent change
  Total Cholesterol | -39.9 [-42.1 to -37.7] | -32.8 [-35.8 to -29.7] | -24.4 [-27.9 to -21.0]
  Triglycerides | -25.3 [-36.0 to -14.6] | -18.8 [-29.8 to -7.8] | -12.0 [-21.3 to -2.7]
  High-Density Lipoprotein Cholesterol (HDL-C) | 10.3 [6.1 to 14.5] | 7.4 [3.7 to 11.0] | 9.9 [3.6 to 16.2]
  Non-HDL-C | -50.1 [-52.7 to -47.6] | -41.4 [-44.8 to -37.9] | -31.3 [-35.4 to -27.1]
  High Sensitivity C-reactive Protein (Hs-CRP) | 73.0 [-84.4 to 230.4] | -2.9 [-36.3 to 30.4] | -13.6 [-39.7 to 12.6]

ADVERSE EVENTS:
Description: Randomized participants
Arm/Group | Ezetimibe + Atorvastatin | Atorvastatin | Rosuvastatin
Serious Adverse Events (participants affected / at risk) | 4/47 | 1/46 | 0/32
Other Adverse Events (participants affected / at risk) | 13/47 | 5/46 | 9/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe + Atorvastatin (N=47) | Atorvastatin (N=46) | Rosuvastatin (N=32)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Heat illness (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Carcinoid tumour of the gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe + Atorvastatin (N=47) | Atorvastatin (N=46) | Rosuvastatin (N=32)
Nasopharyngitis (Infections and infestations) | 7 (8) | 5 (6) | 3 (4)
Blood creatine phosphokinase increased (Investigations) | 3 (4) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish/present any interim results of the study without Sponsor's prior written consent. The investigator further agrees to provide to the sponsor 45 days prior to submission, review copies of abstracts/manuscripts that report any study results. The sponsor has the right to review and comment. If the parties disagree, investigator agrees to meet with the sponsor for the purpose of making good faith efforts to discuss and resolve any such issues or disagreement.